CLINICAL TRIAL: NCT03744260
Title: The Effect of Medial Branch Radiofrequency Ablation on Functional Spinal Stability and Lumbar Multifidi Muscle Architecture Assessed by Magnetic Resonance Imaging and Ultrasound Imaging
Brief Title: Medial Branch Radiofrequency Ablation and Lumbar Multifidi
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Clark Smith, Associate Professor of Rehabilitation and Regenerative Medicine, Columbia University
Other Study IDs: AAAR1440
Record Dates: First submitted 2018-11-14; First posted 2018-11-16 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Spondylosis; Osteoarthritis
Keywords: Lower back pain; Radiofrequency ablation; Spine
MeSH Terms: conditions — Spondylosis; Osteoarthritis; Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Patients undergo ultrasound and lumbar MRI — Patients undergo ultrasound, physical therapy exam and MRI before and after the radiofrequency ablation procedure that they are getting as part of their regular care.

SUMMARY:
The purpose of this study is to evaluate the effects of lumbar medial branch radiofrequency ablation (RFA) on lumbar multifidi muscle size and clinical spinal stability. Specifically, this study is designed to highlight the comparison of multifidi muscle architecture using ultrasound imaging (USI) and MRI before and after lumbar medial branch RFA. This study will also include a commonly utilized functional assessment of the lumbar spine to evaluate the effects of RFA on lumbar spinal stability.

DETAILED DESCRIPTION:
Radiofrequency ablation (RFA) for the lumbar spine (lower back) is a procedure used to treat lower back pain secondary to facet arthritis. The procedure ablates (burns) a small nerve that goes to the arthritic joint in the back. This nerve also innervates a muscle called the multifidus, thought to be important for lumbar stability. The investigators are conducting a study to evaluate if RFA has any impact on multifidi size, spinal stability, and overall function. The tools the investigators will be using to assess the multifidi muscles are musculoskeletal ultrasound, MRI, physical therapy assessment, and functional questionnaires. The goal of the study is to determine if RFA impacts the multifidi in a clinically significant fashion, causing atrophy, spinal instability, and/or functional decline.

ELIGIBILITY:
Inclusion criteria are:

* Aged over 18 years
* Presence of lumbar spondylosis or facet arthropathy (as determined by a radiologist) *Unilateral back pain without radicular symptoms
* Positive physical findings for facet mediated pain (pain with lumbar extension and rotation to affected side)
* Ability to complete outcome measure forms.

Exclusion criteria are:

* Prior spinal surgery
* Prior RFA procedures
* Pregnancy
* Contraindications to MRI
* Presence of therapeutic anti-coagulation, medical co-morbidities that would interfere with the ability to perform the procedure safely
* Presence of neurologic changes
* Active tobacco smoking history
* Presence of active litigation
* Presence of open workers compensation case

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with back pain caused by osteoarthritis or degeneration of the facet joint.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Percentage Change in Volume of multifidus muscle on MRI | Up to 3 months after radiofrequency ablation procedure
  Analysis will include volumetric measurements of the multifidi as well as volumetric assessments of the muscle with fat subtracted.
Percentage Change in Cross Sectional Area of Multifidi | Up to 3 months after radiofrequency ablation procedure
  Area will be measured by MRI scan.

SECONDARY OUTCOMES:
Score on Numeric Pain Rating Scale (NPRS) | Up to 3 months after radiofrequency ablation procedure
  The Numeric Pain Rating Scale (NPRS) is a unidimensional measure of pain intensity in adults. Respondents are asked to select a whole number (0-10 integers) that best reflects the intensity of his/her pain. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
Percentage Score on the Modified Oswestry Disability Index | Up to 3 months after radiofrequency ablation procedure
  This is a patient-completed questionnaire which gives a subjective percentage score of level of function (disability) in activities of daily living in those rehabilitating from low back pain. It examines perceived level of disability in 10 everyday activities of daily living, which each statement scored from 0 (no disability) to 5 (worst pain). An aggregate score (percentage) is then calculated, with 0% indicating no disability to 100%, indicating crippled or bed-bound.

CONTACTS AND LOCATIONS:
Overall Officials: Clark C. Smith, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Vagelos College of Physicians and Surgeons, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No